CLINICAL TRIAL: NCT03657433
Title: Intravenous Infusions of Ferumoxytol Compared to Oral Ferrous Sulfate for the Treatment of Anemia in Pregnancy: A Randomized Controlled Trial
Brief Title: Intravenous Infusions of Ferumoxytol Compared to Oral Ferrous Sulfate for the Treatment of Anemia in Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Meghan Hill, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1807765944
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Iron Deficiency Anemia of Pregnancy
MeSH Terms: interventions — ferrous sulfate; Ferrosoferric Oxide

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferumoxyltol (Experimental): Patients will receive two infusions of Ferumoxyltol, 510mg, intravenously, one week apart.
  Iron studies will be completed at study inclusion and again at presentation for delivery. Cord blood will also be assessed for iron studies.
  Interventions: Drug: Ferumoxytol
- Ferrous Sulfate (Active Comparator): Patients will be provided with oral ferrous sulphate, 325mg, to take 2x daily at home.
  Iron studies will be completed at study inclusion and again at presentation for delivery. Cord blood will also be assessed for iron studies.
  Interventions: Dietary Supplement: Ferrous sulfate 325mg

INTERVENTIONS:
Dietary Supplement: Ferrous sulfate 325mg — Oral tablets supplied for home use
  Arms: Ferrous Sulfate
Drug: Ferumoxytol — Ferumoxytol will be administered in two infusions, one week apart
  Arms: Ferumoxyltol

SUMMARY:
This randomized controlled trial includes pregnant women with anemia. They are randomized to IV iron infusions or to oral iron supplementation. Pregnancy outcomes are assessed.

DETAILED DESCRIPTION:
This is a randomized controlled trial aimed at assessing whether IV Iron administration (Ferumoxytol x 2 infusions) is superior to oral ferrous sulfate for the treatment of iron-deficiency anemia in pregnancy.

140 patients will be randomized in a 1:1 ratio. Patients in the IV Iron group will receive two infusions of Ferumoxytol, one week apart. Patients in the oral Ferrous Sulfate group will receive medication to take at home during their pregnancy.

Patients will have iron studies performed at study entry, and again at presentation for delivery. Cord blood will also be sampled for iron studies.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age >/= 18
* Singleton gestation
* >/=20 weeks gestation, <37 weeks gestation
* Hemoglobin <11g/dL and/or hematocrit <33%
* Able to read/speak English or Spanish

Exclusion Criteria:

* Maternal age <18
* Multiple gestation
* <20 weeks gestation, </= 37 weeks gestation
* Hemoglobin >/=11g/dL and/or hematocrit >/=33%
* Unable to read or speak English or Spanish
* Incarcerated patients

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 124 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin | 1 day - 22 weeks
  We will assess the increase in maternal hemoglobin during the study timeframe

SECONDARY OUTCOMES:
Change in other laboratory values | 1 day - 22 weeks
  Including hematocrit, serum iron, transferrin saturation, ferritin
Blood loss at delivery | 1 day - 22 weeks
  Estimated or quantified blood loss at delivery
Hemoglobin change after delivery | 1 day - 22 weeks
  Measured change in hemoglobin after delivery
Blood transfusion | 1 day - 22 weeks
  Whether the mother requires a blood transfusion
Iron infusion | 1 day - 22 weeks
  Whether the mother requires additional iron infusions
Concentration of substances in cord blood (iron studies) | 1 day - 22 weeks
  Cord blood indices for iron, transferrin saturation and ferritin
Preterm delivery | 1 day - 22 weeks
  Whether the delivery occurs at less than 37 weeks of gestation
Indication for delivery | 1 day - 22 weeks
  Indication for delivery if not spontaneous
Birth weight | 1 day - 22 weeks
  Neonatal weight immediately after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Awomolo AM, McWhirter A, Sadler LC, Coppola LM, Hill MG. Neonatal outcomes from a randomized controlled trial of maternal treatment of iron deficiency anemia with intravenous ferumoxytol vs oral ferrous sulfate. Am J Obstet Gynecol MFM. 2023 Sep;5(9):101063. doi: 10.1016/j.ajogmf.2023.101063. Epub 2023 Jun 20. PMID 37348817
- [Derived] Awomolo AM, McWhirter A, Sadler LC, Coppola LM, Hill MG. Intravenous infusions of ferumoxytol compared to oral ferrous sulfate for the treatment of anemia in pregnancy: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Sep;5(9):101064. doi: 10.1016/j.ajogmf.2023.101064. Epub 2023 Jun 20. PMID 37348816